CLINICAL TRIAL: NCT01792739
Title: The Impact of Lactobacillus Preparation on the Incidence of Diarrhea in Intensive Care Unit-admitted Patients : Randomized Controlled Trial
Brief Title: Lactobacillus Preparation on the Incidence of Diarrhea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ICU_probiotics
Record Dates: First submitted 2012-02-09; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Diarrhea; Death; Pneumonia
Keywords: Probiotics; Diarrhea; Intentive care units
MeSH Terms: conditions — Diarrhea; Death; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kadit B (Experimental): Probiotic Lactobacillus casei variety rhamnosus granules
  Interventions: Drug: Lactobacillus casei variety rhamnosus granules
- Kadit A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus casei variety rhamnosus granules — Lactobacillus casei variety rhamnosus granules
  : 3 gram per day (1g-1g-1g, 3 times per day)
  Other Names: RAMNOS GRANULS
  Arms: Kadit B
Drug: Placebo — Placebo granules
  : 3 gram per day (1g-1g-1g, 3 times per day)
  Arms: Kadit A

SUMMARY:
The purpose of this trial is to clarify the impact of lactobacillus preparation on the incidence of diarrhea in ICU-admitted patients.

Almost all patients in ICU are treated with antibiotics for the effective control of various infections. However, antibiotics-associated diarrhea is another matter of concern. Many previous studies were proved that the use of probiotic lactobacillus preparation can reduce antibiotics-associated diarrhea in ward-admitted patients. In this study, we are planning to perform a similar study in severely ill patients in ICU.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in intensive care unit
* Age more than 19

Exclusion Criteria:

* Diarrhea occurence within 1 week of ICU admission
* Recent history of probiotics use (within 1 month)
* GI obstruction
* History of abnormal symptoms and sign for the probiotics use (rash, edema, sepsis, etc.)
* immunocompromized patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Diarrhea-free days | Duration from the first-administration day of probiotics till the first onset day of diarrhea during ICU residence (up to 8 weeks)
  If patients admit to ICU, the patient can be registered to probiotics or placebo arm. After the registration, probiotics would be administered to the patients. If loose stool >600ml/day occurs during ICU residence, we can determine that occurence of diarrhea.
  "Diarrhea-free days" mean the duration from the day of 1st administration of probiotics till the day of 1st diarrhea.
  If patients are transferred to ward, this study ends in each patient.

SECONDARY OUTCOMES:
28day-mortality | 28 day
  Mortality in 28th day of ICU residence
Positive results of C.difficile toxin | The first onset of diarrhea during ICU residence (up to 8 weeks)
  If diarrhea (>600ml/day) occurs during ICU residence, we will perform C.difficile toxin assays to determine the cause of diarrhea.
ICU-acquired pneumonia | The first day of occurence of ICU-acquired pneumonia (up to 8 weeks)
  Definition of ICU-acquired pneumonia
  1. Newly developed pneumonia during ICU residence
  2. Aggravation of pneumonia during ICU residence

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hoon Lee, Doctor, Principal Investigator — Seoul National University College of Medicine
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam, Bundang-Gu
  - Myongji Hospital, Goyang, Deokyang-gu
  - SMG-SNU Boramae Medical Center, Seoul, Dongjak-gu

REFERENCES:
- [Result] Hickson M, D'Souza AL, Muthu N, Rogers TR, Want S, Rajkumar C, Bulpitt CJ. Use of probiotic Lactobacillus preparation to prevent diarrhoea associated with antibiotics: randomised double blind placebo controlled trial. BMJ. 2007 Jul 14;335(7610):80. doi: 10.1136/bmj.39231.599815.55. Epub 2007 Jun 29. PMID 17604300